CLINICAL TRIAL: NCT00227591
Title: A Phase II Study of Lenalidomide (CC-5013) in Combination With Prednisone for the Treatment of Myelofibrosis With Myeloid Metaplasia
Brief Title: Lenalidomide and Prednisone in Treating Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02976; NCI-2012-02976 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E4903; E4903 (Other: Eastern Cooperative Oncology Group); E4903 (Other: CTEP); U10CA021115 (NIH)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2012-12

CONDITIONS: Essential Thrombocythemia; Polycythemia Vera; Primary Myelofibrosis
MeSH Terms: conditions — Thrombocythemia, Essential; Polycythemia Vera; Primary Myelofibrosis | interventions — Lenalidomide; Prednisone

ARMS (1):
- Treatment (lenalidomide, prednisone) (Experimental): For courses 1 and 2, patients receive oral lenalidomide once daily and oral prednisone once daily on days 1-28. For course 3, patients receive oral lenalidomide once daily on days 1-28 and oral prednisone once on days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, and 27. Patients with stable or responding disease after course 3 receive oral lenalidomide alone once daily on days 1-28 for courses 4-6. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: lenalidomide; Drug: prednisone; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lenalidomide — Given orally (PO)
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well giving lenalidomide together with prednisone works in treating patients with myelofibrosis. Lenalidomide may stop the growth of myelofibrosis by blocking blood flow to the cancer. It may also stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as prednisone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with prednisone may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the rate of complete or partial remission from treatment with a combination of lenalidomide and prednisone in patients with myelofibrosis with myeloid metaplasia.

SECONDARY OBJECTIVES:

I. To examine drug toxicity. II. To examine duration of response. III. To examine the effect of treatment on bone marrow fibrosis, angiogenesis, and cytogenetics.

OUTLINE:

For courses 1 and 2, patients receive oral lenalidomide once daily and oral prednisone once daily on days 1-28. For course 3, patients receive oral lenalidomide once daily on days 1-28 and oral prednisone once on days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25, and 27. Patients with stable or responding disease after course 3 receive oral lenalidomide alone once daily on days 1-28 for courses 4-6. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year and then every 6 months for up to 5 years from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be diagnosed with myelofibrosis with myeloid metaplasia (MMM); agnogenic myeloid metaplasia, post-polycythemic myeloid metaplasia, or post-thrombocythemic myeloid metaplasia are included

  * NOTE: Diagnosis must be confirmed by central pathology review; diagnostic samples must be submitted; patient may register and begin treatment based on the local pathology review. If the central review does not confirm patient's eligibility to participate in the trial, protocol treatment must be discontinued
* Patient must have discontinued chemotherapy (hydroxyurea, alpha interferon, anagrelide, other myelosuppressive agents, thalidomide, or any other experimental therapy) as well as growth factors and systemic use of corticosteroids >= 28 days prior to starting study drug

  * All non-hematologic toxicity must be resolved to =< grade 1
* Patient must be lenalidomide-naïve (never treated with lenalidomide)
* ECOG performance status (PS) of 0, 1, or 2 at study entry
* Hemoglobin level =< 10 g/dL or transfusion-dependent
* Absolute neutrophil count >= 1,000 uL
* Platelet count >= 100,000 uL
* Serum creatinine =< 2.0 mg/dL
* Total bilirubin =< 2.0 mg/dL (if elevated; direct bilirubin =< 2.0 mg/dL)
* AST (SGOT) =< 3 x ULN unless attributed to hepatic extramedullary hematopoiesis
* Women must not be pregnant or breastfeeding because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenetic effects on the developing fetus and newborn are unknown; women of childbearing potential who are sexually active, must use 2 accepted methods of birth control at the same time for 4 weeks prior to lenalidomide treatment, during lenalidomide treatment, and up to 4 weeks after lenalidomide treatment is finished; sexually active males must use a latex condom for contraception during the study and up to 4 weeks after treatment with lenalidomide has ended

  * All females of childbearing potential must have a blood test 10-14 days prior to the start of lenalidomide treatment to rule out pregnancy; another blood test to rule out pregnancy must be done 24 hours prior to the start of treatment with lenalidomide
* Patient must not have any condition, including the presence of laboratory abnormalities, which, based on the physician's opinion, places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Patient must not have any known hypersensitivity to thalidomide or lenalidomide
* Patient must not have any known positive status for HIV or infectious hepatitis type A, B or C
* Patient must not have any other active malignancy

  * NOTE: SWOG patients are strongly encouraged to be registered on SWOG-9007 ("Cytogenetic Studies in Leukemia Patients"); SWOG institutions registering patients to SWOG-9007 should follow the instructions for specimen submission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayalew Tefferi, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Mesa RA, Yao X, Cripe LD, Li CY, Litzow M, Paietta E, Rowe JM, Tefferi A, Tallman MS. Lenalidomide and prednisone for myelofibrosis: Eastern Cooperative Oncology Group (ECOG) phase 2 trial E4903. Blood. 2010 Nov 25;116(22):4436-8. doi: 10.1182/blood-2010-05-287417. Epub 2010 Jul 22. PMID 20651074

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study accrued 48 cases between December 2, 2005 and March 9, 2007. Per two-stage design, the study was suspended on May 31, 2006 for a toxicity and response analysis. Since more than 4 patients achieved a response, the study was reactivated on December 5, 2006. Accrual continued to a total of 48 patients and terminated on March 9, 2007.
Groups:
- Lenalidomide: Lenalidomide 10 mg/day plus prednisone X 28 days X 3 cycles
Period: Overall Study
Arm/Group | Lenalidomide
Started | 48 (48 pts registered to the study)
Began Treatment | 47
Completed | 47
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Response was evaluated for Anemia and Spleen:
  Major anemia response: hemoglobin increase to within normal limits in the absence of transfusion. Minor anemia response: hemoglobin improvement of at least 2 grams per deciliter independent of transfusion support, or achievement of transfusion independence in transfusion-dependent patients. Major spleen response: normalization of spleen size to the range of 12-14 centimeters by ultrasound. Minor spleen response: a 50% or more decrease in excess spleen size by ultrasound. Complete remission (CR): complete resolution of disease-related symptoms, splenomegaly, normalization of peripheral blood count, white cell differential and smear, and normalization of bone marrow histology. Partial remission (PR): a major or minor response in anemia or splenomegaly. Overall Response (OR)=CR + PR, assessed among eligible, treated patients.
Time Frame: Assessed at the end of cycle 3
Population: 6 ineligible patients were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 42
Proportion of participants | 0.26 [0.14 to 0.42]

ADVERSE EVENTS:
Time Frame: During treatment (up to 6 months) and for 30 days after the end of treatment.
Arm/Group | Lenalidomide
Serious Adverse Events (participants affected / at risk) | 47/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=47)
ALT Increased (Metabolism and nutrition disorders) | 1
Abdomen pain (Gastrointestinal disorders) | 1
Alkaline Phosphatase Increased (Metabolism and nutrition disorders) | 1
Anemia (Blood and lymphatic system disorders) | 21
Atrial fibrillation (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bilirubin Increased (Metabolism and nutrition disorders) | 2
Diarrhea without prior colostomy (Gastrointestinal disorders) | 1
Dizziness (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Edema limb (Vascular disorders) | 1
Fatigue (General disorders) | 3
Heart block sick sinus syndrome (Cardiac disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Infection with gr3-4 neutrophils (Infections and infestations) | 1
Leukopenia (Blood and lymphatic system disorders) | 14
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 21
Pain NOS (General disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Pulmonary hypertension (Cardiac disorders) | 1
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 9
Thrombosis (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=47)
AST increased (Metabolism and nutrition disorders) | 8
Anemia (Blood and lymphatic system disorders) | 43
Anorexia (Metabolism and nutrition disorders) | 6
Bilirubin Increased (Metabolism and nutrition disorders) | 8
Constipation (Gastrointestinal disorders) | 10
Diarrhea witout prior colostomy (Gastrointestinal disorders) | 21
Dizziness (General disorders) | 9
Dyspepsia muco (Gastrointestinal disorders) | 8
Edema limb (Vascular disorders) | 15
Extremity limb pain (Musculoskeletal and connective tissue disorders) | 7
Fatigue (General disorders) | 19
Headache (General disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hypokalemia (Metabolism and nutrition disorders) | 8
Insomnia (General disorders) | 8
Leukopenia (Blood and lymphatic system disorders) | 29
Neutropenia (Blood and lymphatic system disorders) | 22
Pain NOS (General disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 9
Sweating (General disorders) | 6
Taste disturbance (General disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 27
Weight loss (General disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less